CLINICAL TRIAL: NCT03372226
Title: Computer-based Self-Help Program for People With Gambling Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neustart
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Gambling, Pathologic
Keywords: Gambling; Problematic Gambling; Pathological Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: The study is a randomly controlled study with 2 conditions: Condition 1: Online Intervention Program (treatment of emotional and gambling-related symptoms), condition 2: Wait-list control group (access to the online program after the post-assessment).
  Two assessments-points, the intervention period (pre-post) is eight weeks. At both measuring points sociodemographic and pathological data are obtained with an internet survey on Unipark®.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online self-help program (Experimental): The intervention group receives the login data for the online program directly following the baseline assessment. The program consists of 10 modules with many interactional exercises and homework-sheets.
  Themes that are addressed in the online-program are for example self-esteem, sleep hygiene, problem solving strategies, mindfulness-based relaxation and attention exercises as well as gambling-specific topics such as money/debt management and impulse control. In addition, the user learns to modify negative and gambling-specific thought distortions, to integrate positive activities into his/her daily routine, strategies to deal with the urge to play as well as ways to regulate debts and to prevent relapse.
  Interventions: Behavioral: Online self-help program
- Wait-list control group (No Intervention): The participants of the wait-list control condition do not receive any new intervention during the intervention period of 8 weeks, but may continue any treatment that has already been started before, including medication. Participants in the wait-list control condition receive full access to the program after completion of the post-assessment.

INTERVENTIONS:
Behavioral: Online self-help program — The program consists of 10 modules with many interactional exercises and homework-sheets. Themes that are addressed in the online-program are for example self-esteem, sleep hygiene, problem solving strategies, mindfulness-based relaxation and attention exercises as well as gambling-specific topics such as money/debt management and impulse control. In addition, the user learns to modify negative and gambling-specific thought distortions, to integrate positive activities into his/her daily routine, strategies to deal with the urge to play as well as ways to regulate debts and to prevent relapse.
  Other Names: Neustart
  Arms: Online self-help program

SUMMARY:
The study examines the effectiveness of a computer-based self-help-program for individuals with problematic or pathological gambling behavior.The main objective of the study is to investigate the extent to which the online program leads to a significant reduction in pathological gambling (primary outcome), depression and gambling-specific dysfunctional thoughts. The program is expected to lead to a significant reduction regarding all measures when compared to a control group. The study is conducted as a randomized-controlled trial with one intervention group and one wait-list control group.

DETAILED DESCRIPTION:
The study examines the effectiveness of a computer-based self-help-program for individuals with problematic and pathological gambling behavior. The main objective of the study is to investigate the extent to which the online program leads to a significant reduction in pathological gambling. The primary outcome is the PG-Y-BOCS as a measure of the severity of pathological gambling symptoms. Secondary outcomes are rates of depression, measured with the PHQ-9 as well as gambling-specific cognitive biases, measured with the GABS. The program is expected to lead to a significant reduction in problematic/pathological gambling behavior (PG-Y-BOCS) and also to declines in both depressive symptoms (PHQ-9) and gambling-specific cognitive biases (GABS). The study is conducted as a randomized-controlled trial with one intervention group and one wait-list control group. The intervention group receives the login data directly following the baseline survey and can use the program over a period of 8 weeks, whereas the wait-list control group receives access to the program after completion of the post-survey.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* access to internet
* adequate usage of German language
* willingness to participate in two short (25-30 minutes) online surveys
* willingness to use the online program over a period of 8 weeks (participants that do not use the program are also included in the analysis)
* willingness to leave an (anonymous) email-address
* existence of the wish to receive treatment

Exclusion Criteria:

* existence of a lifetime diagnosis of schizophrenia or bipolar disorder
* existence of an acute suicidal tendency (assessed with item 9 of the PHQ-9, ≥3)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Pathological Gambling Adaptation of Yale-Brown Obsessive Compulsive Scale (PG-Y-BOCS) | 1 week
  The total score consists of ten items that measure the severity of gambling symptoms within the past week. The first five questions assess urges and thoughts associated with gambling, whereas the last five questions assess the behavioral component of the disorder. The sum score of each subscale ranges from 0-20. Each subscale can be analyzed separately as well as together as a total score (primary outcome). The total score can be interpreted as follows: 0-7 sub-clinical, 8-15 mild, 16-23 moderate, 24-31 severe and 32-40 extreme gambling symptoms.

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 depression module (PHQ-9) | 1 week
  The Patient Health Questionnaire - 9 depression module is a self-rating measure of depressive symptom severity. The psychometric properties of the PHQ-9 are very good, with high internal consistency (Cronbach's α = .86 - .89; Kroenke, Spitzer, & Williams, 2001). Its sum score ranges from 0 to 27, with scores from 0-4 indicating minimal depression, 5-9 mild depression, 10-14 moderate depression and 15-27 severe depression.
Gambling Attitudes and Beliefs Survey (GABS) | time of assessment
  The GABS is a self-report questionnaire which explores gambling-related dysfunctional beliefs. In this study, we use a 15-item version of the GABS. Responses can be given on a four-point Likert scale (from 'strongly agree' to 'strongly disagree').
South Oaks Gambling Screen (SOGS) | 6 months
  20-items self-report measure to screen for engagement in gambling activities and gambling-related problems. A score between 0-2 corresponds to non-problematic gambling, a score of 3-4 to at-risk gambling, and a score of 5-20 to probable pathological gambling.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Gehlenborg J, Moritz S, Bucker L. The Dimensional Structure of the Gambling Attitudes and Beliefs Survey: Challenging the Assumption of the Unidimensionality of Gambling-Specific Cognitive Distortions. J Gambl Stud. 2023 Mar;39(1):75-86. doi: 10.1007/s10899-022-10133-7. Epub 2022 May 28. PMID 35633435
- [Derived] Bucker L, Gehlenborg J, Moritz S, Westermann S. A randomized controlled trial on a self-guided Internet-based intervention for gambling problems. Sci Rep. 2021 Jun 22;11(1):13033. doi: 10.1038/s41598-021-92242-8. PMID 34158553
- [Derived] Bucker L, Westermann S, Kuhn S, Moritz S. A self-guided Internet-based intervention for individuals with gambling problems: study protocol for a randomized controlled trial. Trials. 2019 Jan 23;20(1):74. doi: 10.1186/s13063-019-3176-z. PMID 30674348